CLINICAL TRIAL: NCT03282136
Title: Incretin Treatment and Combined to SGLT2i Effect in Type 2 Diabetes Mellitus Patients Affected by Heart Failure With Depressed Ejection Fraction, and Treated by Cardiac Resynchronization Therapy With a Defibrillator.
Brief Title: SGLT2i and Incretin and CRTd.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, principal investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Campania
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure | interventions — Incretins; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- incretin arm (Active Comparator): T2DM with HF treated by CRTd participants will be assigned prospectively to an intervention (incretin therapy plus conventional hypoglycemic drug therapy) according to study protocol to evaluate the effect of the drug on cardiac deaths, all cause deaths, and hospital admission for heart failure.
  Interventions: Drug: Incretin Effect; Device: Cardiac Resynchronization therapy defibrillator device
- conventional hypoglycemic drug arm (Placebo Comparator): T2DM with HF treated by CRTd participants will be assigned prospectively to SGLT2i therapy (plus conventional hypoglycemic drug therapy) according to study protocol to evaluate the effect of the drug on cardiac deaths, all cause deaths, and hospital admission for heart failure.
  Interventions: Device: Cardiac Resynchronization therapy defibrillator device
- Incretin added to SGLT2i (Active Comparator): T2DM with HF treated by CRTd participants will be assigned prospectively to SGLT2i added to incretin therapy (plus conventional hypoglycemic drug therapy) according to study protocol to evaluate the effect of the drug on cardiac deaths, all cause deaths, and hospital admission for heart failure.
  Interventions: Drug: SGLT-2 inhibitor

INTERVENTIONS:
Drug: Incretin Effect — The patients will receive incretins therapy.
  Arms: incretin arm
Device: Cardiac Resynchronization therapy defibrillator device — The patients will receive a Cardiac Resynchronization therapy defibrillator device
  Arms: conventional hypoglycemic drug arm; incretin arm
Drug: SGLT-2 inhibitor — The patients will receive SGLT2i therapy.
  Arms: Incretin added to SGLT2i

SUMMARY:
Incretin therapy and sodium-glucose- transporter2 inhibitors (SGLT2i) are a treatment for type 2 diabetes (T2DM) affected by heart failure (HF) and treated with cardiac resynchromization therapy (CRT). In this study the investigators will recruit T2DM patients affected by HF with depressed ejection fraction and treated by CRT. These patients will randomly be treated by incretin v/s SGLT2i vs combined therapy with incretin+SGLT2i (and added to conventional hypoglicemic drugs). In these patients investigators will report at follow up CRT-d responders rate, mortality, and hospital admission for HF worsening. Combined therapy with incretin and SGLT2i may reduce hospital admissions for HF in T2DM v/s incretin and/or SGLT2i therapy (added to conventional hypoglicemic drugs).

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years, with clinical hystory of T2DM non insulin dependent, and diagnosed failing heart with depressed ejection fraction; CRTd recipients.

Exclusion Criteria:

* T2DM in insuline therapy; renal impairment, chronic inflammatory and systemic diseases; neoplastic diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality, and cardiac cause mortality. | 12 months
CRT responders | 12 months

SECONDARY OUTCOMES:
hospital admissions for HF | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sardu C, Paolisso P, Sacra C, Santamaria M, de Lucia C, Ruocco A, Mauro C, Paolisso G, Rizzo MR, Barbieri M, Marfella R. Cardiac resynchronization therapy with a defibrillator (CRTd) in failing heart patients with type 2 diabetes mellitus and treated by glucagon-like peptide 1 receptor agonists (GLP-1 RA) therapy vs. conventional hypoglycemic drugs: arrhythmic burden, hospitalizations for heart failure, and CRTd responders rate. Cardiovasc Diabetol. 2018 Oct 22;17(1):137. doi: 10.1186/s12933-018-0778-9. PMID 30348145